CLINICAL TRIAL: NCT04459975
Title: Acute Kidney Injury and Renal Outcomes for COVID-19 Patients in Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CoV-AKI_2020
Record Dates: First submitted 2020-06-12; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: on Occurrence of Acurate Kidney Injury During Intensive Care Unit; Abnormalities of Urinary Analysis
Keywords: Acurate Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI (-): patients treated in ICU for COVID-19 infection and without occurrence of AKI (define as creatinine > 1,5x baseline according with KDIGO guidelines)
- AKI (+): patient treated in ICU for COVID-19 infection and with occurrence of AKI among which:
  • Severe AKI patients (define as creatinine > 3x baseline or need for renal replacement therapy according with KDIGO guidelines) who will participate to biocollection and to post-mortem biopsy (if death).
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Comorbidities, creatinine levels, urinary analysis, hemodynamic, respiratory status, co-medication will be collected from medical files for each patient.
  Specific datas from patients with AKI will be collected from medical files For severe acute patients, serum and urinary analysis will performed to identify the underlying cause of kidney injury For severe AKI patients who will die, post-mortem renal biopsy will be performed, for histopathological analysis
  Groups: AKI (+)

SUMMARY:
The actual COVID-19 epidemy is an unprecedented healthcare problem. Although acute respiratory distress syndrome is the main organ failure, acute kidney injury (AKI) has appeared to be more frequent and more severe than expected. Some data suggested a potential direct renal tropism of the virus, or undirect injury by "cytokine storm".

The aims of this study are:

1. To describe incidence, severity and mortality associated with AKI during covid-19 infection in ICU
2. To identify specific risk factors for AKI
3. To explore pathophysiologic mechanism of AKI during COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection (by qRT-PCR and/or TDM typical lesion)
* Needing intensive care

Exclusion Criteria:

* End Stage Renal Disease patients (with pre-existent dialysis)
* Intensive care support for less than 72h (transfer in conventional unit or death)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients supported in intensive care units for covid-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the incidence, the severity and the mortality associated with AKI during COVID-19 severe infection | 7 months
  AKI will be defined according with KDIGO guidelines: increase in creatinine of more than 1,5 fold compared to baseline Severe CVOID-19 infection is defined as 1/ confirm COVID-19 infection (by TDM and/or qRT-PCR) 2/ Requirement of ICU support during more than 72h

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive care units attached to the Hospices Civils de Lyon (HCL), Lyon, France